CLINICAL TRIAL: NCT03372876
Title: Protein Intake Immediately After Resistance Exercise Does Not Promote Additional Increase on Lean Mass, Strength and Functional Capacity in Postmenopausal Women: a Randomized Clinical Trial
Brief Title: Protein Timing, Lean Mass, Strength and Functional Capacity Gains in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Erick Prado de Oliveira, PhD, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2.023.127
Record Dates: First submitted 2017-12-10; First posted 2017-12-14 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Proteins; Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein-carbohydrate (PC) (protein intake after exercise) (Experimental): ingested 30 g of whey protein immediately after exercise and 30 g of maltodextrin in the afternoon. The resistance exercise was performed equally by both groups.
  Interventions: Dietary Supplement: Protein and carbohydrate supplementation
- Carbohydrate-protein (CP) (protein intake far to exercise) (Placebo Comparator): ingested 30 g of maltodextrin immediately after exercise and 30 g of whey protein in the afternoon. The resistance exercise was performed equally by both groups.
  Interventions: Dietary Supplement: Protein and carbohydrate supplementation

INTERVENTIONS:
Dietary Supplement: Protein and carbohydrate supplementation — Participants were randomly assigned to protein-carbohydrate group (PC) (n=17), that ingested 30 g of whey protein immediately after exercise and 30 g of maltodextrin in the afternoon; and to carbohydrate-protein group (CP) (n=17), that ingested 30 g of maltodextrin immediately after exercise and 30 g of whey protein in the afternoon. Both groups performed the same resistance training protocol in the morning, 3 times a week, at 70% of 1-maximum repetition (1-RM) during 8 weeks.
  Other Names: Resistance exercise

SUMMARY:
This study evaluated the effect of protein intake immediately after resistance exercise on lean mass, strength, and functional capacity gains in postmenopausal women. Participants were randomly assigned to protein-carbohydrate group (PC) (n=17), that ingested 30 g of whey protein immediately after exercise and 30 g of maltodextrin in the afternoon; and to carbohydrate-protein group (CP) (n=17), that ingested 30 g of maltodextrin immediately after exercise and 30 g of whey protein in the afternoon. Both groups performed the same resistance training protocol in the morning.

DETAILED DESCRIPTION:
Both groups performed the same training protocol, differing only the time of protein or carbohydrate supplementation. The dietary assessment was made through the 24-hour food recall, being conducted at the beginning, middle and end of the intervention. Resistance exercises for upper and lower limbs will be performed, at 70% of one repetition maximum. One maximum repetition (1-RM), handgrip strength and 1-mile walk were performed.

ELIGIBILITY:
Inclusion Criteria:

* Women in the postmenopausal period (menopausal for at least one year, confirmed by laboratory diagnostic tests menopause - LH and high FSH and estradiol decreased);
* Healthy;
* Who agree to participate and sign the consent term.

Exclusion Criteria:

* The one who does not provide the necessary information for the development of the study;
* Present orthopedic limitations;
* Patients with previously diagnosed and treatment of diseases such as type II diabetes mellitus, hypertension and cardiovascular disease.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
Changes in the lean mass of postmenopausal women practicing resistance exercise | Before and immediately after the intervention (initial moment and 8 weeks after start of the intervention)

SECONDARY OUTCOMES:
Changes on strength of postmenopausal women practicing resistance exercise | Before and immediately after the intervention (initial moment and 8 weeks after start of the intervention)
Changes on functional capacity of postmenopausal women practicing resistance exercise | Before and immediately after the intervention (initial moment and 8 weeks after start of the intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Erick P. de Oliveira, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Branco FMS, Carneiro MAS, Rossato LT, Nahas PC, Teixeira KRC, de Oliveira GN Jr, Orsatti FL, de Oliveira EP. Protein timing has no effect on lean mass, strength and functional capacity gains induced by resistance exercise in postmenopausal women: A randomized clinical trial. Clin Nutr. 2020 Jan;39(1):57-66. doi: 10.1016/j.clnu.2019.01.008. Epub 2019 Jan 17. PMID 30691866